CLINICAL TRIAL: NCT02792387
Title: Some Characteristics of Interaction Between Heart and Kidneys in Cardio-Renal Syndrome Type 1 and Type 2
Brief Title: The Role of CVP and EF in Patients With Cardio-renal Syndromes
Acronym: RoCVPinCRSs
Status: Completed | Type: Observational
Sponsor: Tbilisi State University (Other)
Responsible Party: Principal Investigator, George Lobzhanidze, MD, Tbilisi State University
Other Study IDs: TSU100
Record Dates: First submitted 2016-05-16; First posted 2016-06-07 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure
Keywords: cardio-renal syndrome; right heart dysfunction; central venous pressure; eGFR; low-flow theory
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Central Venous Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: CVP measurement — CVP measurements had been performed with an electronic pressure transducer in spontaneously breathing non-ventilated patients. Central vein access was established trough the subclavian or internal jugular veins. Mean CVP was recorded for each patient, measured in mmHg.

SUMMARY:
The aim of the study is to explore association between increased central venous pressure, Ejection Fraction and renal dysfunction (eGFR) in patients with Cardio-Renal Syndromes type 1 and 2. The pilot study was set to provide the expected correlation coefficient for a sample size determination of the subsequent study.

DETAILED DESCRIPTION:
OBJECTIVES

The aim of the study is to explore association between increased central venous pressure (CVP), Ejection Fraction (EF) and renal dysfunction (eGFR) in patients with Cardio-Renal Syndromes type 1 and 2.

BACKGROUND

The pathophysiology of impaired renal function in cardiovascular disease is multifactorial. Recent investigations suggest that management of patients based on low-flow theory does not lead to improved outcomes. Relative importance of right heart dysfunction (manifested as increased CVP) has not been evaluated . Precise understanding of bidirectional pathways by which the heart and kidneys influence each other is necessary to define optimal treatment strategies specific to the subtypes, as therapies directed towards one organ system may have beneficial or unfavorable effects on the other.

METHODS

The study is of non-experimental (observational) type, based on retrospective chart review. The patients' personal identifiers are concealed and an anonymized datasets used (unique code given to each patient, which is kept secure under the control of hospital staff).

ELIGIBILITY:
Inclusion Criteria:

* HF (NYHA class I - IV, with preserved and reduced EF) and reduced GFR (Cardio-Renal Syndromes 1 and 2)

Exclusion Criteria:

* Independent risk factors for renal impairment (e.g. diabetes, sepsis)
* Primary nephropathy or secondary nephropathy due to diseases other than HF

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent in-patient treatment at medical centers
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
renal impairment (defined as a Glomerular Filtration Rate less than 60 mL/min per 1.73 m2) | through study completion, an average of 1 year
  Estimated Glomerular Filtration Rate has been assessed with the Modification of Diet in Renal Disease formula

CONTACTS AND LOCATIONS:
Overall Officials: George Lobzhanidze, MD, Principal Investigator — Tbilisi State University

IPD SHARING:
Plan to Share IPD: No